CLINICAL TRIAL: NCT05723016
Title: Serum Anti-Müllerian Hormone Levels and Its Association With Aneuploidy Rates in Human Blastocysts
Brief Title: Anti-Müllerian Hormone and Embryo Aneuploidy
Status: Completed | Type: Observational
Sponsor: Clinica de la Mujer Medicina Reproductiva, Chile (Other)
Responsible Party: Principal Investigator, Jose Antonio Moreno, MD, PhD, Clinica de la Mujer Medicina Reproductiva, Chile
Other Study IDs: AMH 2023
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Infertility; Aneuploidy
Keywords: AMH; IVF; Aneuploidy; PGT-a; anti-mullerian hormone; oocyte quality
MeSH Terms: conditions — Infertility; Aneuploidy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- AMH < 0.5 ng/ml
  Interventions: Other: preimplantation genetic test for aneuploidies (PGT-a)
- AMH 0.5-0.99 ng/ml
  Interventions: Other: preimplantation genetic test for aneuploidies (PGT-a)
- AMH 1.0-1.49 ng/ml
  Interventions: Other: preimplantation genetic test for aneuploidies (PGT-a)
- AMH 1.5-1.99 ng/ml
  Interventions: Other: preimplantation genetic test for aneuploidies (PGT-a)
- AMH 2.0-4.99 ng/ml
  Interventions: Other: preimplantation genetic test for aneuploidies (PGT-a)
- AMH > 5.0 ng/ml
  Interventions: Other: preimplantation genetic test for aneuploidies (PGT-a)

INTERVENTIONS:
Other: preimplantation genetic test for aneuploidies (PGT-a) — preimplantation genetic test for embryo aneuploidies after IVF

SUMMARY:
The goal of this observational study is to determine is there an association between the rates of aneuploidy and the different ranges of serum Antimullerian hormone (AMH) levels.

Retrospective, single-centre study of patients undergoing IVF and preimplantation genetic testing with aneuploidy at the blastocyst stage between January 2018 and December 2022.

ELIGIBILITY:
Inclusion Criteria:

* All started cycles planned to be followed by preimplantation genetic testing for aneuploidies (PGT-A). PGT-A is proposed to the couples for the following reasons: advanced maternal age, recurrent miscarriage, repeated implantation failure or severe male infertility factor; it is also offered to all patients with a good prognosis who desired information regarding the ploidy status of their embryos.

Exclusion Criteria:

* Data from oocyte donation cycles

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Patients who underwent a first IVF cycle with PGT-A at the blastocyst stage
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Aneuplody rate | 4 years

SECONDARY OUTCOMES:
Clinical pregnancy rate | 4 years
Miscarriage rate | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica de la Mujer Medicina Reproductiva, Viña del Mar, Región de Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: Undecided